CLINICAL TRIAL: NCT00330746
Title: Randomized Phase II Study of Cetuximab in Combination With Gemcitabine or Gemcitabine Followed by Cetuximab in Advanced Non Small-cell Lung Cancer Patients Who Are Not Candidates for Platinum Based Therapy.
Brief Title: CALC-1 (Cetuximab in Advanced Lung Cancer): Study of 2 Methods of Combining Cetuximab and Gemcitabine in Patients With Advanced Non Small-cell Lung Cancer
Acronym: CALC-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALC-1; 2004-002811-98 (EudraCT Number)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: elderly; chemotherapy; targeted therapy; combination therapy; sequential therapy; randomized phase II; one year survival
MeSH Terms: interventions — Cetuximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): cetuximab and gemcitabine combination
  Interventions: Drug: cetuximab; Drug: gemcitabine
- B (Experimental): gemcitabine followed by cetuximab (sequential)
  Interventions: Drug: gemcitabine; Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — 400 mg/m2 first dose then weekly at 250 mg/m2 until disease progression
  Arms: A
Drug: gemcitabine — 1200 mg/m2 days 1 and 8 every 3 weeks for a maximum of 6 cycles
  Arms: A
Drug: gemcitabine — 1200 mg/m2 IV days 1 and 8 every 3 weeks for a maximum of 6 cycles
  Arms: B
Drug: cetuximab — 400 mg/m2 first dose followed by 250 mg/m2 weekly
  Arms: B

SUMMARY:
The purpose of this study is to select the more promising method of combining cetuximab with gemcitabine for treating patients with advanced non small-cell lung cancer, who are not candidates for platinum based therapy.

DETAILED DESCRIPTION:
The standard treatment for advanced non small cell lung cancer (NSCLC) is combination chemotherapy with cisplatin or carboplatin. Due to its toxicity, this therapy may not be suited for certain patients including the elderly, those whose general condition is poor. Combining chemotherapy with a biologic agent ("targeted therapy") is a new strategy being evaluated for the treatment of NSCLC, and cetuximab is one of the drugs that has shown promise for its activity and tolerability. This study aims to determine the more promising of 2 methods of combining gemcitabine with cetuximab (in combination vs. sequential administration), in two groups of patients who are not candidates for combination platinum based chemotherapy: patients under age 70 with performance status 2 (expected enrollment 42) , and patients over age 70 (expected enrollment 58).

Patients will be randomly assigned to one of two treatment arms:

* Arm A: Cetuximab + Gemcitabine:

  * Cetuximab given intravenously weekly AND
  * Gemcitabine given intravenously for a maximum of 6 cycles (on days 1 and 8 of each 3 week cycle)
* Arm B: Gemcitabine followed by Cetuximab:

  * Gemcitabine given intravenously for a maximum of 6 cycles (on days 1 and 8 of each 3 week cycle) THEN
  * Cetuximab given intravenously weekly

In Arm B, Cetuximab is administered as maintenance therapy when there has been an objective response to chemotherapy, or as second line therapy in patients who had disease progression during chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age > 18
* Histological diagnosis of non small-cell lung cancer (NSCLC)
* Stage III B or Stage IV disease
* Contraindications to platinum based therapy (age > 70 or age < 70 with ECOG performance status 2)
* At least one site of metastasis (target or non-target)
* Life expectancy of at least 3 months
* ECOG <3
* Neutrophils > 1500/mm3, platelets > 100,000/mm3, hemoglobin > 9g/dl
* Bilirubin < 1.5 x the upper normal limit
* SGOT and SGPT < 2.5 x the upper normal limits (< 5 x the upper normal limit in the presence of hepatic metastasis)
* Creatinine < 1.5 x the upper normal limit
* Adequate method of contraception (male and female), when there is risk of conception.

Exclusion Criteria:

* Symptomatic cerebral metastasis
* Previous chemotherapy for advanced disease
* Adjuvant chemotherapy within the previous 6 months
* Radiation therapy within previous 4 weeks
* Any experimental drug therapy within the previous 4 weeks
* Previous exposure to monoclonal antibodies, signal transduction inhibitors or EGFR targeting therapy
* Clinically relevant cardiopathy or myocardial infarct within the last 12 months
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease
* Known allergy to one or more of the experimental treatments
* Known alcohol or substance abuse
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or give informed consent
* Pregnant or breastfeeding females
* History of malignant neoplasm within the previous 5 years (not including non-melanoma skin carcinoma and in-situ carcinoma of the uterine cervix, provided they are being adequately treated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
one year survival rate | one year

SECONDARY OUTCOMES:
toxicity | weekly
overall survival | 18 months
overall response rate | one year
prognostic role of cetuximab associated skin toxicities | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — S.G. Moscati Hopital, Avellino, Italy, Division of Medical Oncology; Fortunato Ciardiello, M.D., Ph.D, Principal Investigator — Second Univesity of Naples, Italy; Chair Medical Oncology; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; Ciro Gallo, M.D., Ph.D, Principal Investigator — Second University of Naples, Italy; Chair of Medical Statistics
Locations (25):
- Italy (25):
  - Azienda Sanitaria S. Giuseppe Moscati, Monteforte Irpino, AV
  - Ospedale A. Cardarelli, Campobasso, CB
  - Università di Chieti, Chieti, CH
  - Ospedale Umberto di Frosinone, Frosinone, FR
  - Ospedale Villa Scassi, Genova, GE
  - Ospedale di Gaeta, Gaeta, LT
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina, ME
  - Ospedale S. Giuseppe, Milan, MI
  - Istituto Scientifico S. Raffaele, Milan, MI
  - Ospedale S. Paolo, Milan, MI
  - Ospedale S. Gerado, Monza, MI
  - Azienda Ospedaliera C. Poma, Mantova, MN
  - Policlinico Giaccone, Palermo, PA
  - Ospedale di Prato, Prato, PO
  - Ospedale S. Croce, Fano, PS
  - Ospedale S. Salvatore, Pesaro, PU
  - Ospedale Civile Umberto I, Nocera Inferiore, SA
  - Azienda Ospedaliera Universitaria Senese, Siena, SI
  - Ospedale E. Morelli, Sondalo, SO
  - Presidio Ospedaliaro Alto Gardo e Ledro, Arco, TN
  - Ospedale S. Chiara, Trento, TN
  - Azienda Ospedaliera Di Busto Arsizio, Saronno, VA
  - Divisione di Oncologia Medica, U.S.L.L. 13, Noale, VE
  - Azienda Ospedaliera Cardarelli, Napoli
  - Second University of Naples, Napoli

REFERENCES:
- [Result] Gridelli D, Mencoboni M, Carrozza F, Viganò MG, Gebbia V, Verusio C, Maione P, Gallo C, Perrone F, Ciardiello F. Cetuximab (C) and gemcitabine (G) in elderly or adult PS2 advanced non small-cell lung cancer (NSCLC) patients (pts): The CALC1 randomised phase II trials. Journal of Clinical Oncology 26: 2008 (May 20 suppl; abstr 8117)
- [Result] Gridelli C, Morabito A, Gebbia V, Mencoboni M, Carrozza F, Vigano MG, Verusio C, Bollina R, Mattioli R, Valerio MR, Valmadre G, Maione P, Rossi A, Cascone T, Morgillo F, Di Maio M, Piccirillo MC, Gallo C, Perrone F, Ciardiello F. Cetuximab and gemcitabine in elderly or adult PS2 patients with advanced non-small-cell lung cancer: The cetuximab in advanced lung cancer (CALC1-E and CALC1-PS2) randomized phase II trials. Lung Cancer. 2010 Jan;67(1):86-92. doi: 10.1016/j.lungcan.2009.03.021. PMID 19380175